CLINICAL TRIAL: NCT01342536
Title: A Culturally Adapted Depression Intervention for African American Adults
Brief Title: African American Depression Intervention Trial (AADI)
Acronym: AADI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0109, 2011-0234; R01MD005905-01A1 (NIH)
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Coping Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lifestyle counseling (OHDC) (Experimental): Oh Happy Day Class (OHDC) is a culturally-specific, 12-week cognitive behavioral group counseling intervention designed for African American adults experiencing depression
  Interventions: Behavioral: Coping with Depression Course (CWD) and Oh Happy Day Class (OHDC)
- lifestyle counseling (CWD) (Active Comparator): Coping with Depression Course (CWD) is a 8-week cognitive behavioral group counseling depression intervention
  Interventions: Behavioral: Coping with Depression Course (CWD) and Oh Happy Day Class (OHDC)

INTERVENTIONS:
Behavioral: Coping with Depression Course (CWD) and Oh Happy Day Class (OHDC) — The OHDC is a culturally adapted, cognitive behavioral group counseling intervention. The OHDC is theoretically grounded in social learning theory and an Afrocentric paradigm (Nguzo Saba). It uses a social support group and psychoeducation format so participants learn skills to help them in coping and reducing symptoms of depression. The OHDC is offered over 13 weeks with 2-hour sessions in a clinical setting.
  The CWD, an evidence-based cognitive behavioral depression intervention. The CWD is offered over 8 weeks with 2-hour sessions in a clinical.
  Arms: lifestyle counseling (OHDC), lifestyle counseling (CWD)

SUMMARY:
Primary Aim 1: Examine effectiveness of the Oh Happy Day Class (OHDC) compared to the Coping With Depression (CWD)in increasing retention, adherence, engagement, satisfaction, and treatment-seeking. The investigators hypothesize the OHDC compared to the CWD will result in greater increases in: 1a. retention, 1b. adherence, 1c. engagement, and 1d. satisfaction at the middle and end of the intervention, and 2.e. greater increase in treatment-seeking 3-, 6-, 9-, and 12- months post-intervention. Outcome measures: logs: attendance, homework completion, class-participation level; Client Satisfaction Inventory; and Cornell Service Index. Primary Aim 2: Examine effectiveness of the OHDC in reducing symptoms of depression at the middle and immediate end of the intervention, and 3-, 6-, 9-, and 12- months post-intervention. The investigators hypothesize the OHDC will result in greater reduction in depressive symptoms compared to the CWD at 3-months post-intervention. Outcome measures: Center for Epidemiologic Studies Depression Scale and Quick Inventory of Depression Symptoms. Secondary Aim 3: Examine the effectiveness of the OHDC in improving self-reports of mental and physical health status and reducing self-reports of perceived disability. The investigators hypothesize the OHDC compared to the CWD will result in greater self-report of: 3a. improved mental and physical health status, and 3b. reduced self-report of disability at the immediate end of the intervention and 3-,6-, 9-, 12- months post-intervention. Outcome measures: SF-12 Health Survey, and World Health Organization Disability Assessment Schedule.

Public Health Impact: Based on CAI research, the OHDC has the potential to be four times more effective than the CWD. If our hypotheses are proven, the OHDC will be the first evidence-based culturally adapted depression intervention designed specifically for African American men and women between the ages of 30-60.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria. Self-identified African-American men and women, between the ages of 30 to 60, with symptoms of depression as evidenced by data from the Composite International Diagnostic Interview 2.1 (CIDI). Although age of inclusion is broad, our pilot studies have shown positive outcomes with mixed aged groups

Exclusion Criteria:

* Exclusion criteria. Individuals will be excluded from the study if they have: (1) self-reported alcohol or other drug abuse/dependence, (2) major psychotic illnesses, such as schizophrenia as evidenced by results of the CIDI, (3) self-reported changes in antidepressants (dosage or type) less than 6 weeks prior to participating in the study, (4) self-report of current psychotherapy treatment, or (5) self-report of current suicidal ideations (our psychiatrist will conduct additional suicide risk assessment and facilitate referral for appropriate care.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2011-12-14 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D) | up to 4 years
  Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D scale is a 20-item self-report inventory developed by NIMH to assess the frequency and severity of depression symptoms in the past week. Respondents indicate how often each symptom was experienced during the past week on a four-point scale from "Rarely or none of the time (0)", "Some or a little of the time (1)", "Occasionally or a moderate amount of the time (2)", or "Most or all of the time (3)". Item scores are summed for analyses, with a possible range 0-60. A standard cutoff score of 16 indicates depressive symptoms.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology (QIDS) | up to 4 years
  The 16-item Quick Inventory of Depressive Symptomatology (QIDS) using DSM-IV criteria assesses depressive symptom severity and symptom change. The QIDS has a clinician-rated and self-report format. Studies show high internal consistency for the QIDS-CR (0.85) and QIDS-SR(0.86). Scores range from 0-27 and higher scores suggest higher severity. The QIDS also has high concurrent validity with the SF-12.

CONTACTS AND LOCATIONS:
Overall Officials: Earlise C Ward, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Mental Health Center of Dane County, Madison, Wisconsin
  - Milwaukee Health Services, INC, Milwaukee, Wisconsin